## Combining Treatment Components in Transdiagnostic Therapy for Anxiety and Depression: A Randomized Controlled Trial

Date: May 13th, 2024

## Statistical analysis plan

An overview of measures at each time point is provided in Table 1. Multilevel models will be employed as the primary analytic model, where time (level 1) is nested within individuals (level 2). Models will include a random intercept in addition to random slope if it improves model fit. For the covariance between the intercept and slope, a variance component and unstructured pattern will be tested. We will first evaluate the respective efficacy of each treatment component compared to no treatment (i.e., waiting period) and then compare the efficacy of the two treatment components when delivered first. For our primary analysis, we will compare potential sequencing effects in a time (pre-treatment through post-treatment) x group (mindful emotion awareness first vs. cognitive flexibility first) interaction analysis. Finally, we will explore the potential maintenance of effect at follow-up and at this point compare the two arms. The number of individuals who experience reliable clinical change in each of the groups will also be compared (Jacobson & Truax, 1991). Demographic and clinical baseline characteristics will be explored as moderators.

**Table 1.** Overview of measures at each time point

| | Baseline (T1) | Pre-treatment (T2) | Mid-treatment<br>(T3) | Post-treatment | Follow-up (T5) | Session<br>(Ts1-6) |
|---|---|---|---|---|---|---|
| | | | | (T4) | | |
| Primary outcomes | | | | | | |
| PHQ-9 | X | X | X | X | X | X |
| BAI | X | X | X | X | X | X |
| GAD-7 | X | X | X | X | X | |
| SIAS | X | X | X | X | X | |
| PDSS-SR | X | X | X | X | X | |
| Secondary outcomes | | | | | | |
| WHO-5 | X | X | X | X | X | |
| RRS brooding subscale | X | X | X | X | X | X |
| PSWQ | X | X | X | X | X | |
| AWS | | | | | | X |
| EQ decentering subscale | X | X | X | X | X | Xa |
| ERQ reappraisal subscale | X | X | X | X | X | X |
| FFMQ-15 | X | X | X | X | X | X |
| PDQ-D | X | X | X | X | X | |
| Treatment specific variables | | | | | | |
| Experience of therapy | | | | X | X | X |
| WAI-SR | | | | | | $X^b$ |
| IO | | | | | | X |
| Clinical evaluation | | | | | | |
| ADIS-5 | X | | | | | |
| WAIS-IV Digit span | X | | | | | |
| TMT-A | X | | | | | |
| TMT-B | X | | | | | |
| COWAT | X | | | | | |
| WAIS-IV Coding | X | | | | | |
| STROOP | X | | | | | |
| WAIS-IV Information | X | | | | | |

Notes. Abbreviations: ADIS-5 = The Anxiety and Related Disorders Interview Schedule for DSM-5 (Brown & Barlow, 2014), AWS = the Ambulatory Worry Scale (Kramer et al., 2021), BAI = Beck's Anxiety Inventory (Beck et al., 1988; Beck & Steer, 1991), COWAT = Controlled Oral Word Association Test (Harrison et al., 2000), EQ = The Experiences Questionnaire (Fresco et al., 2007), ERQ = Emotion Regulation Questionnaire (Gross & John, 2003), FFMQ-15 = Five Facet Mindfulness Questionnaire – 15 (Baer et al., 2006),

GAD-7 = General Anxiety Disorder-7 (Spitzer et al., 2006), IO = Information Overload scale (adapted from Jensen et al., 2014; see Appendix E), PDQ-D = Perceived Deficits Questionnaire – Depression (Fehnel et al., 2016), PDSS-SR = the Panic Disorder Severity Scale – Self-Report Version (Houck et al., 2002), PHQ-9 = Patient Health Questionnaire-9 (Kroenke et al., 2001; Spitzer et al., 1999; Spitzer et al., 2000), PSWQ = The Penn State Worry Questionnaire (Meyer et al., 1990), RRS = The Ruminative Response Scale (Treynor et al., 2003), SIAS = the Social Interaction Anxiety Scale (Mattick & Clarke, 1998), TMT = Trail Making Test (Reitan, 1958), WAI-SR = Working Alliance Inventory – Short Revised (Munder et al., 2010), WAIS-IV = Wechsler Adult Intelligence Scale – Fourth Edition (Wechsler, 2008), STROOP = The Stroop Color and Word Test (Stroop, 1935), WHO-5 = the World Health Organization-5 questionnaire (Bech, 1999; Topp et al., 2015).

- a: A brief version reduced to 5 items (cf. O'Toole et al., 2019) is used in the session questionnaires.
- b: Only included in Ts2 and Ts5.

## References

- Baer, R. A., Smith, G. T., Hopkins, J., Krietemeyer, J., & Toney, L. (2006). Using Self-Report Assessment Methods to Explore Facets of Mindfulness. *Assessment*, 13(1), 27-45. https://doi.org/10.1177/1073191105283504
- Bech, P. (1999). Health-related quality of life measurements in the assessment of pain clinic results. *Acta Anaesthesiologica Scandinavica*, *43*(9), 893-896. https://doi.org/10.1034/j.1399-6576.1999.430906.x
- Beck, A. T., Epstein, N., Brown, G., & Steer, R. A. (1988). An inventory for measuring clinical anxiety: psychometric properties. *Journal of Consulting and Clinical Psychology*, 56(6), 893-897. https://doi.org/10.1037//0022-006x.56.6.893
- Beck, A. T., & Steer, R. A. (1991). Relationship between the beck anxiety inventory and the Hamilton anxiety rating scale with anxious outpatients. *Journal of Anxiety Disorders*, 5(3), 213-223. https://doi.org/https://doi.org/10.1016/0887-6185(91)90002-B
- Brown, T. A., & Barlow, D. H. (2014). *Anxiety and Related Disorders Interview Schedule for DSM-5, adult and lifetime version: clinician manual.* Oxford University Press.
- Fehnel, S. E., Forsyth, B. H., DiBenedetti, D. B., Danchenko, N., François, C., & Brevig, T. (2016). Patient-centered assessment of cognitive symptoms of depression. *CNS Spectrums*, 21(1), 43-52. https://doi.org/10.1017/s1092852913000643
- Fresco, D. M., Moore, M. T., van Dulmen, M. H., Segal, Z. V., Ma, S. H., Teasdale, J. D., & Williams, J. M. (2007). Initial psychometric properties of the experiences questionnaire: validation of a self-report measure of decentering. *Behavior Therapy*, 38(3), 234-246. https://doi.org/10.1016/j.beth.2006.08.003
- Gross, J. J., & John, O. P. (2003). Individual Differences in Two Emotion Regulation Processes: Implications for Affect, Relationships, and Well-Being. *Journal of personality and social psychology*, 85(2), 348-362. <a href="https://doi.org/10.1037/0022-3514.85.2.348">https://doi.org/10.1037/0022-3514.85.2.348</a>
- Harrison, J. E., Buxton, P., Husain, M., & Wise, R. (2000). Short test of semantic and phonological fluency: normal performance, validity and test-retest reliability. *British Journal of Clinical Psychology*, 39(2), 181-191. https://doi.org/10.1348/014466500163202
- Houck, P. R., Spiegel, D. A., Shear, M. K., & Rucci, P. (2002). Reliability of the self-report version of the panic disorder severity scale. *Depression and anxiety*, 15(4), 183-185. https://doi.org/10.1002/da.10049
- Jacobson, N. S., & Truax, P. (1991). Clinical significance: A statistical approach to defining meaningful change in psychotherapy research. *Journal of Consulting and Clinical Psychology*, *59*(1), 12-19. https://doi.org/10.1037/0022-006X.59.1.12
- Jensen, J. D., Carcioppolo, N., King, A. J., Scherr, C. L., Jones, C. L., & Niederdieppe, J. (2014). The cancer information overload (CIO) scale: establishing predictive and discriminant validity. *Patient Education and Counseling*, 94(1), 90-96. <a href="https://doi.org/10.1016/j.pec.2013.09.016">https://doi.org/10.1016/j.pec.2013.09.016</a>
- Kramer, A. C., Neubauer, A. B., Leonhardt, A., Brose, A., Dirk, J., & Schmiedek, F. (2021). Ambulatory assessment of rumination and worry: Capturing perseverative cognitions in children's daily life. *Psychological assessment*, 33(9), 827-842. https://doi.org/10.1037/pas0001020
- Kroenke, K., Spitzer, R. L., & Williams, J. B. (2001). The PHQ-9: validity of a brief depression severity measure. *Journal of General Internal Medicine*, 16(9), 606-613. <a href="https://doi.org/10.1046/j.1525-1497.2001.016009606.x">https://doi.org/10.1046/j.1525-1497.2001.016009606.x</a>
- Mattick, R. P., & Clarke, J. C. (1998). Development and validation of measures of social phobia scrutiny fear and social interaction anxiety. *Behaviour research and therapy*, *36*(4), 455-470. <a href="https://doi.org/10.1016/s0005-7967(97)10031-6">https://doi.org/10.1016/s0005-7967(97)10031-6</a>

- Meyer, T. J., Miller, M. L., Metzger, R. L., & Borkovec, T. D. (1990). Development and validation of the Penn State Worry Questionnaire. *Behaviour research and therapy*, 28(6), 487-495. https://doi.org/10.1016/0005-7967(90)90135-6
- Munder, T., Wilmers, F., Leonhart, R., Linster, H. W., & Barth, J. (2010). Working Alliance Inventory-Short Revised (WAI-SR): psychometric properties in outpatients and inpatients. *Clinical psychology and psychotherapy*, 17(3), 231-239. <a href="https://doi.org/10.1002/cpp.658">https://doi.org/10.1002/cpp.658</a>
- O'Toole, M. S., Renna, M. E., Mennin, D. S., & Fresco, D. M. (2019). Changes in Decentering and Reappraisal Temporally Precede Symptom Reduction During Emotion Regulation Therapy for Generalized Anxiety Disorder With and Without Co-Occurring Depression. *Behavior Therapy*, 50(6), 1042-1052. https://doi.org/10.1016/j.beth.2018.12.005
- Reitan, R. M. (1958). Validity of the Trail Making Test as an Indicator of Organic Brain Damage. *Perceptual and Motor Skills*, 8(3), 271-276. https://doi.org/10.2466/pms.1958.8.3.271
- Spitzer, R. L., Kroenke, K., Williams, J. B., & Löwe, B. (2006). A brief measure for assessing generalized anxiety disorder: the GAD-7. *Arch Intern Med*, *166*(10), 1092-1097. https://doi.org/10.1001/archinte.166.10.1092
- Spitzer, R. L., Kroenke, K., Williams, J. B., & the Patient Health Questionnaire Primary Care Study Group. (1999). Validation and Utility of a Self-report Version of PRIME-MD: The PHQ Primary Care Study. *Jama*, 282(18), 1737-1744. https://doi.org/10.1001/jama.282.18.1737
- Spitzer, R. L., Williams, J. B., Kroenke, K., Hornyak, R., & McMurray, J. (2000). Validity and utility of the PRIME-MD patient health questionnaire in assessment of 3000 obstetric-gynecologic patients: the PRIME-MD Patient Health Questionnaire Obstetrics-Gynecology Study. *American Journal of Obstetrics and Gynecology*, 183(3), 759-769. <a href="https://doi.org/10.1067/mob.2000.106580">https://doi.org/10.1067/mob.2000.106580</a>
- Stroop, J. R. (1935). Studies of interference in serial verbal reactions. *Journal of experimental psychology*, *18*(6), 643-662. <a href="https://doi.org/10.1037/h0054651">https://doi.org/10.1037/h0054651</a>
- Topp, C. W., Østergaard, S. D., Søndergaard, S., & Bech, P. (2015). The WHO-5 Well-Being Index: A Systematic Review of the Literature. *Psychotherapy and psychosomatics*, 84(3), 167-176. https://doi.org/10.1159/000376585
- Treynor, W., Gonzalez, R., & Nolen-Hoeksema, S. (2003). Rumination Reconsidered: A Psychometric Analysis. *Cognitive Therapy and Research*, 27(3), 247-259. https://doi.org/10.1023/A:1023910315561
- Wechsler, D. (2008). Wechsler Adult Intelligence Scale Fourth Edition (WAIS-IV). Pearson. <a href="https://www.pearsonassessments.com/store/usassessments/en/Store/Professional-Assessments/Cognition-%26-Neuro/Wechsler-Adult-Intelligence-Scale-%7C-Fourth-Edition/p/100000392.html">https://www.pearsonassessments.com/store/usassessments/en/Store/Professional-Assessments/Cognition-%26-Neuro/Wechsler-Adult-Intelligence-Scale-%7C-Fourth-Edition/p/100000392.html</a>